CLINICAL TRIAL: NCT02856867
Title: Nintedanib Plus mFOLFOX6 for Previously Untreated Metastatic Esophagogastric Adenocarcinoma (MEGAN): A Randomized, Placebo-controlled, Triple-blind Phase II Study
Brief Title: Nintedanib Plus mFOLFOX6 for Previously Untreated Metastatic Esophagogastric Adenocarcinoma (MEGAN)
Acronym: MEGAN
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC-1418-GITCG; 2016-002361-58 (EudraCT Number)
Record Dates: First submitted 2016-07-28; First posted 2016-08-05 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Esophagogastric Adenocarcinoma; Metastatic Disease; No Previous Chemotherapy for Metastatic Esophagogastric Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — nintedanib; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- mFOLFOX6 + Nintedanib (Active Comparator): Patients will receive nintedanib in combination with mFOLFOX6 (5-Fluorouracil 400 mg/m2 bolus on day 1, 5-Fluorouracil 2400 mg/m2 continuous infusion over 46 hours starting on day 1, Leucovorin 400 mg/m2 on day 1, Oxaliplatin 85 mg/m2 on day 1) via IV infusions every 2 weeks (14 days).
  Dose modification of nintedanib and mFOLFOX6 is allowed. Patients may continue to receive protocol therapy as long as they have not experienced any adverse events requiring permanent discontinuation of study medication and have not demonstrated disease progression.
  Interventions: Drug: Nintedanib; Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- mFOLFOX6 + Placebo (Placebo Comparator): Patients will receive placebo in combination with mFOLFOX6 (5-Fluorouracil 400 mg/m2 bolus on day 1, 5-Fluorouracil 2400 mg/m2 continuous infusion over 46 hours starting on day 1, Leucovorin 400 mg/m2 on day 1, Oxaliplatin 85 mg/m2 on day 1) via IV infusions every 2 weeks (14 days).
  Dose modification of placebo and mFOLFOX6 is allowed. Patients may continue to receive protocol therapy as long as they have not experienced any adverse events requiring permanent discontinuation of study medication and have not demonstrated disease progression.
  Interventions: Drug: Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Placebo

INTERVENTIONS:
Drug: Nintedanib
  Arms: mFOLFOX6 + Nintedanib
Drug: Fluorouracil
Drug: Leucovorin
Drug: Oxaliplatin
Drug: Placebo
  Arms: mFOLFOX6 + Placebo

SUMMARY:
This is a prospective, multicenter, randomized, placebo-controlled, triple-blind phase II trial. The randomization will be a 1:1 randomization (experimental arm:control arm). This study will enroll patients with histologically confirmed esophagogastric adenocarcinoma with metastatic disease. Patients will have had no previous chemotherapy for metastatic esophagogastric cancer. Patients will receive nintedanib or placebo in combination with mFOLFOX6 (5-Fluorouracil 400 mg/m2 bolus on day 1, 5-Fluorouracil 2400 mg/m2 continuous infusion over 46 hours starting on day 1, Leucovorin 400 mg/m2 on day 1, Oxaliplatin 85 mg/m2 on day 1) via IV infusions every 2 weeks (14 days). Dose modification of nintedanib or placebo and mFOLFOX6 is allowed. Patients may continue to receive protocol therapy as long as they have not experienced any adverse events requiring permanent discontinuation of study medication and have not demonstrated disease progression.

The primary objective is to test the hypothesis that progression free survival (PFS) is prolonged in HER2-negative patients with untreated metastatic esophagogastric adenocarcinoma when treated with nintedanib plus modified FOLFOX6 (mFOLFOX6) as compared to placebo plus mFOLFOX6. The analyses will be performed when 124 events for PFS will have been observed in the pooled arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophagogastric adenocarcinoma with metastatic (M1) disease
* HER2-negative tumors as per local assessment (according to Rüschoff-Criteria)
* Presence of at least one evaluable lesion per RECIST v1.1
* Representative formalin fixed, paraffin embedded tumor blocks or unstained tissue slides, either from the primary tumor or a metastatic lesion, must be available for histological central review of FGFR2 and associated oncogenic pathway and tumor stroma analyses
* Age 18 years or older
* ECOG performance status 0-1
* Within 7 days prior to treatment start: adequate bone marrow, liver and renal function and coagulation parameters:

  * Neutrophils ≥ 1.5 x 109/L
  * Hemoglobin ≥ 9 g/dL (or ≥ 5.6 mmol/L). Blood transfusions or the administration of hematopoietic growth factors are allowed to achieve these baseline values
  * Platelets ≥ 100 x 109/L. Platelet transfusions or the administration of hematopoietic growth factors are allowed to achieve these baseline values
  * Bilirubin ≤ 1.5 x ULN
  * Patients with Gilbert syndrome and/or bilirubin <2 ULN and normal AST/ALT are eligible
  * SGPT/ALT and SGOT/AST ≤ 2.5 x ULN for patients with liver metastasis
  * SGPT/ALT and SGOT/ AST ≤ 1.5x ULN for patients without liver metastasis
  * Serum creatinine ≤ 1.5 x ULN or creatinine clearance/eGFR > 45 ml/min assessed as per local standard method
  * No proteinuria CTCAE grade 2 or greater
  * International normalized ratio (INR) < 2, prothrombin
  * Prothrombin time (PT) and partial thromboplastin time (PTT) >50% of institutional ULN.
  * No Child Pugh B or C hepatic impairment
* Women of childbearing potential (WOCP): defined as a sexually mature woman who 1) has not undergone a hysterectomy or bilateral oophorectomy or 2) has not been naturally post-menopausal (amenorrhoea following cancer therapy does not rule out childbearing potential) for at least 12 consecutive months (i.e. has had menses at any time in the preceding 12 consecutive months), must:

  * Have a negative serum pregnancy test within 7 days prior to randomization.
  * Agree to remain sexually abstinent, have a partner who is sterile (i.e., vasectomy), or use two medically effective methods of contraception during dosing and through 90 days after last study treatment. An effective method is the combination of the following (a+b): a. Hormonal method eg, birth control pills; b. Placement of an intrauterine device (IUD) or intrauterine system (fUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/ gel/film/ cream/vaginal suppository. This requirement should be followed from screening through 24 weeks after last study treatment.
  * During treatment: Patient should agree to urine pregnancy test to be performed before each treatment;
  * Agree to discontinue treatment in case of pregnancy or positive pregnancy test.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 6 months after the last study treatment.
* Sexually active male participants must use a barrier method of contraception (e.g., condom).
* Before patient registration/randomization, written informed consent must be obtained according to International Council for Harmonisation/Good Clinical Practice (ICH/GCP) and national/local regulations.

Exclusion Criteria:

* Previous chemotherapy for metastatic esophagogastric cancer (Neoadjuvant or adjuvant systemic treatments have to be finished at least (≥) 6 months before study inclusion)
* History or clinical evidence of central nervous system metastasis or leptomeningeal tumor spread.
* Other malignant disease in the previous 5 years (apart from basal-cell cancer of the skin or pre-invasive cervical cancer).
* Other anti-cancer therapy (systemic therapy, radiotherapy, surgery) within 28 days prior to treatment start and while on protocol treatment.
* Treatment with another investigational agent within 28 days prior to treatment start and while on protocol treatment.
* Chronic diarrhea or short bowel syndrome
* Legal incapacity or limited legal capacity
* Known hypersensitivity to nintedanib
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration/randomization in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12; Primary Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 30 months from first patient in

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years from first patient in
Objective Response Rate (ORR, according to RECIST v1.1) | 30 months from first patient in
Safety and tolerability (adverse event assessment according to CTCAE v 4.0) | 30 months from first patient in
Quality of Life evaluated by questionnaires | 30 months from first patient in
  Quality of life will be evaluated with these two questionnaires:
  * EORTC QLQ-30 version 3.0
  * EORTC QLQ-Life gastric-specific

CONTACTS AND LOCATIONS:
Overall Officials: Maren Knoedler, Study Chair — Universitaetsklinikum Leipzig, Germany